CLINICAL TRIAL: NCT00810914
Title: Patient Controlled Epidural Infusion Vs. Continuous Epidural Infusion: Obstetrical and Neonatal Outcomes
Brief Title: Patient Controlled Epidural Analgesia Versus Continuous Epidural Infusion: Obstetrical and Neonatal Outcomes
Acronym: Epidural
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MemorialCare (Other)
Responsible Party: Michael Haydon, MD, Women's Pavilion at Miller Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 333-06; MHS 801001-R433306
Record Dates: First submitted 2008-02-19; First posted 2008-12-18 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Pain
Keywords: Patient controlled epidural anesthesia; Pain control in labor
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Continuous epidural infusion of medication for method of pain relief
  Interventions: Drug: bupivicaine epidural
- 2 (Experimental): continuous epidural infusion in conjuction with patient controlled anesthesia (PCA)
  Interventions: Drug: bupivicaine epidural infusion patient epidural
- 3 (Experimental): patient controlled anesthesia only this arm has pt controlled medication delivery. (PCA)
  Interventions: Drug: bupivicaine

INTERVENTIONS:
Drug: bupivicaine epidural — bupivicaine continuous epidural infusion
  Other Names: Marcaine
  Arms: 1
Drug: bupivicaine epidural infusion patient epidural — bupivicaine
  Other Names: marcaine
  Arms: 2
Drug: bupivicaine — patient controlled anesthesia only
  Other Names: marcaine
  Arms: 3

SUMMARY:
The investigators intend to perform a large randomized trial using standardized obstetrical and anesthetic practice at a single institution to determine the effects of patient controlled epidural analgesia on obstetrical and neonatal outcomes.

DETAILED DESCRIPTION:
Women in their first pregnancy in spontaneous labor desiring epidural anesthesia will be randomized to one of three groups. Each group will initially be given intrathecal bolus. Before and 30 minutes after the initial bolus, the patient's verbal pain score will be recorded. The continuous epidural infusion group (Group I) will be started immediately on a continuous pump infusion.They will also have the opportunity to give a PCA bolus Finally, the patient controlled epidural group (Group III) will be able to give a bolus every 20 minutes with no continuous infusion. Each group will also be allowed 2 boluses,by the anesthesia staff in the event that their pain is not controlled by the indicated study medication. An hourly evaluation of verbal pain score and maternal mobility will be recorded. After delivery, obstetrical outcomes, neonatal outcomes, anesthesia interventions, and patient satisfaction questionnaires will then be collected.

ELIGIBILITY:
Inclusion Criteria:

* Early labor
* Nulliparous

Exclusion Criteria:

* Inductions
* Breech
* Contraindications to regional anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Total bupivicaine used | End of labor

SECONDARY OUTCOMES:
maternal satisfaction | End of labor

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haydon, MD, Principal Investigator — Memorial care Health Sytem Physcian
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States